CLINICAL TRIAL: NCT05721560
Title: Pre-market Clinical Investigation Inovedis SINEFIX
Brief Title: SINEFIX-2022 Pilot Phase
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: BAAT Medical Products B.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SINEFIX-2022
Record Dates: First submitted 2023-01-17; First posted 2023-02-10 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Rotator Cuff Tears (RCTs)
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Intervention Model Description: Pilot phase: single-arm prospective non-comparative single-centre study phase
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SINEFIX (Experimental): Rotator cuff repair with the SINEFIX implant, using the SINEFIX instruments
  Interventions: Device: Rotator cuff repair with the SINEFIX

INTERVENTIONS:
Device: Rotator cuff repair with the SINEFIX — Treatment of rotator cuff lesions of size up to 2 cm using the SINEFIX implant and instruments

SUMMARY:
Shoulder pain is one of the most commonly reported musculoskeletal complaints, which negatively affects upper limb use, night rest, daily life activities, work, sports performance and autonomy. Rotator cuff disease represents the most common cause of shoulder pain and it is responsible for up to 70% of all shoulder related visits to clinicians. Its incidence furthermore is expected to grow as the population ages. A wide range of conditions are included under the umbrella term of rotator cuff disease, including rotator cuff tendinopathy, subacromial bursal pathology, and partial-thickness or full-thickness rotator cuff tears (RCTs). The latter ones, i.e. rotator cuff tears, form the indications for which the test devices, the SINEFIX implant and instruments, are intended.

Despite the high prevalence of this condition, the pathophysiology and healing potential are not well understood, making the condition challenging to predictably treat in some patient populations. RCTs may occur in young people as a consequence of trauma (e.g. acute shoulder dislocation), however RCTs typically present in middle-aged or elderly people and cannot always be attributed to precipitating events or trauma. Instead, they can be attributed to degenerative processes, and are therefore referred to as degenerative RCTs.

For RCTs, treatment options include both surgical and non-surgical (conservative) procedures.

In this context, the SINEFIX implant and instruments were developed to treat adult patients with rotator cuff lesions of size up to 2 cm through arthroscopic reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Patient indicated for surgical repair of the rotator cuff tear according to current guidelines
* Patient aged 18 years or older
* Up to 2 cm tear size of supraspinatus, infraspinatus (medio-lateral)
* Up to 2 cm tear size of supraspinatus, infraspinatus (anterior-posterior)

Exclusion Criteria:

* Subject has had previous rotator cuff, arthroplasty or fracture procedures on the operative shoulder
* History of alcoholism, drug abuse, psychological or other emotional problems likely to interfere with participation in the study follow-up schedule and assessments
* Inflammatory arthropathies
* Subject with a contraindication/non-compliance for MRI examination
* Subject 's unwillingness to undergo surgical rotator cuff repair, participate in post-operative rehabilitation program, and / or adhere to follow up schedule
* Pregnant and breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2023-09-12 (Actual); Primary Completion 2024-07-23 (Actual); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Healing integrity | 3 months post operation
  Healing integrity will be assessed with the MRI by evaluating the visibility of the tendon underneath the implant (yes/no)
Re-tear rate | 3 months post operation
  Re-tear rate will be assessed with MRI
Dislocation of the implant | 3 months post operation
  Presence of dislocation of the implant will be assessed with MRI (yes/no)
Bursitis | 3 months post operation
  Presence of bursitis will be assessed with MRI (yes/no)

SECONDARY OUTCOMES:
Surgery time | Immediately post procedure
  The total procedure duration will be recorded as the surgery time
Usability and workflow assessment | Immediately post procedure
  Usability and workflow assessment will be evaluated after each intervention through a practitioner's questionnaire covering different aspects of the implant and instruments
Functional and clinical outcome after rotator cuff repair | At 6 months, 1 and 2 years follow-up
  Functional and clinical outcome after rotator cuff repair will be assessed using the total Constant Murley score, which ranges from 0 (worst outcome) to 100 (best outcome)
Functional and clinical outcome after rotator cuff repair as compared with baseline | At 6 months, 1 and 2 years follow-up
  Functional and clinical outcome after rotator cuff repair will be assessed using the change of the total Constant Murley score (range 0-100) as compared to baseline
Shoulder function after rotator cuff repair (subjective evaluation) | At 10 weeks, 6, 12, and 24 months
  Shoulder function after rotator cuff repair (subjective evaluation) will be assessed through the Subjective Shoulder Value (SSV) which ranges from 0% to 100% (best outcome)
Shoulder function after rotator cuff repair (physical examination-active external rotation) | At 10 weeks, 6, 12, and 24 months
  Shoulder function after rotator cuff repair (physical examination) will be assessed through a physical examination with assessment of range of motion for active external rotation (range 0°-90°)
Shoulder function after rotator cuff repair (physical examination-active anteversion) | At 10 weeks, 6, 12, and 24 months
  Shoulder function after rotator cuff repair (physical examination) will be assessed through a physical examination with assessment of range of motion for active anteversion (0°-180°)
Healing integrity | At 6, 12, and 24 months
  Healing integrity will be assessed with the MRI by evaluating the visibility of the tendon underneath the implant (yes/no)
Re-tear rate | At 6, 12, and 24 months
  Re-tear rate will be assessed with MRI
Dislocation of the implant | At 6, 12, and 24 months
  Presence of dislocation will be assessed with MRI (yes/no)
Bursitis | At 6, 12, and 24 months
  Presence of bursitis will be assessed with MRI (yes/no)
Complications | During the follow up time (up to 24 months)
  Complications will be systematically reported. Complications of particular interest for the purpose of the study are neurological problems, bleeding, impaired wound healing, infection and frozen shoulder.
Patient satisfaction | At 10 weeks, 6, 12, 24 months
  The patient will be asked to rate his/her satisfaction with outcome of the surgical repair (0=completely unsatisfied, 1=unsatisfied, 2=satisfied, 3=completely satisfied)
Safety endpoint | During the intervention and the follow up time (up to 24 months)
  Safety of the device will be evaluated by systematically reporting device deficiencies (DDs), adverse events (AEs) and serious adverse events (SAEs) and by monitoring the frequency and incidence of these events

CONTACTS AND LOCATIONS:
Locations (1):
- Orthopädisch Chirurgisches Centrum (OCC), Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No